CLINICAL TRIAL: NCT00966004
Title: Phase III Study of YM178 - A Placebo-controlled, Double-blind, Group Comparison Study in Patients With Overactive Bladder
Brief Title: A Study to Evaluate Safety and Efficacy of YM178 in Patients With Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 178-CL-048
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urge incontinence; YM178; Overactive Bladder; Urgency; Urinary incontinence; mirabegron; Micturition
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence | interventions — mirabegron; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- YM178 group (Experimental): oral
  Interventions: Drug: YM178
- Placebo group (Placebo Comparator): oral
  Interventions: Drug: Placebo
- tolterodine group (Active Comparator): oral
  Interventions: Drug: tolterodine

INTERVENTIONS:
Drug: YM178 — oral
  Other Names: mirabegron
  Arms: YM178 group
Drug: Placebo — oral
  Arms: Placebo group
Drug: tolterodine — oral
  Other Names: Detrol; Detrusitol
  Arms: tolterodine group

SUMMARY:
The purpose of the study is to evaluate the effect of YM178 in patients with overactive bladder for 12-week administration.

DETAILED DESCRIPTION:
This study examines the superiority of YM178 over the placebo and evaluates the safety and pharmacokinetics of YM178 in patients with overactive bladder, and to compare the efficacy and safety of YM178 over those of tolterodine, the control drug, without a non-inferiority test.

The drug administration period is 14 weeks in total, consisting of 2 weeks for placebo (pre-investigation period) and 12 weeks for the investigational drug (treatment period).

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptoms of overactive bladder for at least 24 weeks before initiation of the pre-investigational period
* Patient capable of walking to the lavatory without assistance and measuring the urine volume by him/herself
* Patient with an average frequency of micturition of 8 or more times per 24-hour period
* Written informed consent has been obtained

Exclusion Criteria:

* Patients without experience of urge incontinence before informed consent
* Patients given a clear diagnosis of stress incontinence
* Patients with transient symptoms suspected of overactive bladder (drug induced, psychogenic, etc)
* Patients complicated with urinary tract infection, urinary stones, and/or interstitial cystitis
* Patients with a previous history of recurrent urinary tract infection
* Patients complicated with or with a history of bladder tumor or prostatic tumor
* Patients confirmed to have a post-void residual volume of ≥ 100 mL or with a clinically significant lower urinary tract obstructive disease
* Patients given medication for the treatment of lower urinary tract obstructive disease within 4 weeks before the pre-investigational period
* Patients with an indwelling catheter or practicing intermittent self-catheterization
* Patients given radiotherapy influencing urethral functions, or thermotherapy for benign prostatic hyperplasia
* Patients given surgical therapy which may influence urethral functions within 24 weeks before the pre-investigational period
* Patients with uncontrolled hypertension or with a pulse rate ≥ 110 bpm or < 50 bpm
* Patients with polyuria exceeding 3000 mL in mean daily urine volume
* Patients meeting any of the following in the examinations

  * Patients with abnormal electrocardiogram judged inappropriate as subjects by the ECG Evaluation Committee
  * Patients with AST (GOT) or ALT (GPT) 2.5 times higher than the upper limit of the normal range (or 100 IU/L)
  * Patients with a blood creatinine level ≥ 2.0 mg/dL

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2009-07-24 (Actual); Primary Completion 2010-02-15 (Actual); Study Completion 2010-02-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean number of micturitions per 24 hours | Within a 12-week treatment period

SECONDARY OUTCOMES:
Change from baseline in the mean number of urgency episodes per 24 hours | Within a 12-week treatment period
Change from baseline in the mean number of urinary incontinence episode per 24 hours | Within a 12-week treatment period
Change from baseline in the mean number of urge incontinence episodes per 24 hours | Within a 12-week treatment period
Change from baseline in the mean volume voided per micturition | Within a 12-week treatment period
Change from baseline in mean number of nocturia episodes | Within a 12-week treatment period
Change from baseline in domain score of quality of life scores as assessed by King's health questionnaire | Within a 12-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Chūbu
  - Kantou
  - Kinki
  - Kyushu

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=193